CLINICAL TRIAL: NCT03381963
Title: Hemostatic Profiles Associated With Use of Aromatase Inhibitors and Tamoxifen in Women With Breast Cancer : a Prospective Cohort Study
Brief Title: Hemostatic Profiles of Endocrine Therapies for Breast Cancer
Acronym: HEMOBREAST
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marc Blondon, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2016-119
Record Dates: First submitted 2017-11-05; First posted 2017-12-22 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Breast Neoplasms; Venous Thromboembolism
Keywords: tamoxifen; aromatase inhibitors; breast cancer; venous thromboembolism
MeSH Terms: conditions — Breast Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Aromatase inhibitors
- Tamoxifen

SUMMARY:
The aim of this prospective cohort study is to evaluate the modifications of the biological hemostatic profile associated with the use of endocrine therapy in women with breast cancer (tamoxifen or aromatase inhibitors).

DETAILED DESCRIPTION:
In this cohort study, women with breast cancer and an indication for endocrine therapy will be prospectively enrolled. At the 1st visit (before the start of endocrine therapy (tamoxifen or aromatase inhibitor)) and at the 2nd visit (at ~3 months after the start of treatment), demographical / clinical data and blood samples will be collected. We will evaluate the hemostatic biological profiles associated with the use of endocrine therapy by comparing hemostatic biomarkers before and during its use.

ELIGIBILITY:
Inclusion Criteria: adult women with a diagnosis of non-metastatic breast cancer and an indication for adjuvant endocrine therapy

Exclusion Criteria:

* lack of consent
* planned chemotherapy
* personal history of venous thromboembolism
* ongoing anticoagulant treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a new diagnosis of non-metastatic breast cancer and a planned adjuvant endocrine therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in thrombin generation, including APC sensitivity ratio | three months

SECONDARY OUTCOMES:
Change in levels of coagulation factors | three months
  Levels of the following coagulation factors will be measured and compared before and after use of endocrine treatments: antithrombin, protein C, protein S, D-dimer, fibrinogen, F VII, F VIII
Change in fibrinolytic time | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Blondon M, Bodmer A, Thouvenin L, Lecompte T, Righini M, Fontana P, Casini A. Differential impact of tamoxifen and aromatase inhibitors on thrombin generation: the prospective HEMOBREAST cohort. Blood Adv. 2022 May 10;6(9):2884-2892. doi: 10.1182/bloodadvances.2021006623. PMID 35086148